CLINICAL TRIAL: NCT02592980
Title: Evaluation of a Pharmacogenetic-based Warfarin Dosing Algorithm in Patients With Low Time in Therapeutic Range - Study Design
Brief Title: Evaluation of a Pharmacogenetic-based Warfarin Dosing Algorithm in Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other); Farmoquimica S.A. (Industry); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PF
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional anticoagulation (Experimental): For the Traditional Anticoagulation group, the physician will adjust the dose according to the current INR value based on current guidelines
  Interventions: Drug: Traditional anticoagulation
- Pharmacogenetic anticoagulation (Experimental): For the Pharmacogenetic Anticoagulation group, the dose will be prescribed based on data from each patient applied in a pharmacogenetic algorithm. In some cases, used algorithm may provide a counter-intuitive dose, i.e., a dose that is not adequate for adjusting the current patient' INR (for example, a higher dose for a patient that already has a high INR). In these cases, the physician will adjust the dose following clinical criteria based on published guidelines
  Interventions: Genetic: Pharmacogenetic anticoagulation

INTERVENTIONS:
Genetic: Pharmacogenetic anticoagulation — The investigators use a algorithm pharmacogenetic for adjust only the first dose in the study.
  Other Names: Warfarin
  Arms: Pharmacogenetic anticoagulation
Drug: Traditional anticoagulation — The physician will adjust the dose according to current INR value based on guidelines.
  Other Names: Warfarin
  Arms: Traditional anticoagulation

SUMMARY:
Background: Time in therapeutic range (TTR) is a measurement of quality of warfarin therapy and lower TTR values (<50%) are associated with greater risk of thromboembolic and bleeding events. Recently, the investigators developed a pharmacogenetic-based warfarin dosing algorithm specifically calibrated for a Brazilian patient sample. The newly developed algorithm was shown to be more accurate for individuals from the Brazilian population than algorithms developed from international samples. The aims of this study are: to evaluate the impact of a genetic-based algorithm, compared to traditional anticoagulation, in the time to achieve the therapeutic target and in TTR percentage; and to assess the cost-effectiveness of genotype-guided warfarin dosing in a specific cohort of patients with low TTR (<50%) from a tertiary cardiovascular hospital. Methods/Design: The investigators will recruit 300 patients with TTR<50% based on the last three INR values. At the first consultation, patients will be randomized into two groups: TA (Traditional Anticoagulation) group and PA (Pharmacogenetic Anticoagulation) group. For the first group, the physician will adjust the dose according to current INR value and, for the second group, a pharmacogenetic algorithm will be used. At the second, third, fourth and fifth consultations (with an interval of 7 days each) INR will be measured and, if necessary, the dose will be adjusted based on guidelines. Afterwards, patients who are INR stable will begin measuring their INR in 30 day intervals; if the patient´s INR is not stable, the patient will return in 7 days for a new measurement of the INR. The main outcomes will be the time to achieve the therapeutic target and the percentage of TTR at 4 and 12 weeks. In addition, as a secondary end-point, pharmacoeconomic analysis will be carried out. Discussion: With a sample size of 150 patients for each arm separately, the study will have a power of 93% to observe a difference of 10% between TTR means of the TA and PA groups. This randomized study will include patients with low TTR and it will evaluate whether a population-specific genetic algorithm might be more effective than traditional anticoagulation for a selected group of poorly anticoagulated patients.

DETAILED DESCRIPTION:
Investigators will recruit 300 patients with low TTR (<50%) from the Heart Institute- Clinical Hospital- University of São Paulo Medical School (InCor- HCFMUSP). The patients will be randomized into two groups: Traditional Anticoagulation (TA) group and Pharmacogenetic Anticoagulation (PA) group. The study protocol was approved by the Ethics Committee for Medical Research on Human Beings of the Clinical Hospital of the University of São Paulo Medical School (SDC 4033/14/013). Signed informed consent will be obtained from all participants.

Only patients with atrial fibrillation, above 18 years, and with TTR <50% based on the last three values of INR will be included in this study. Patients will not be included if they have reached a stable dose of warfarin, liver dysfunction, alcoholism, use of another anticoagulant, use of chemotherapy, or if they do not meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with atrial fibrillation, above 18 years, and with TTR <50% based on the last three values of INR will be included in this study.

Exclusion Criteria:

* Patients will not be included if they have reached a stable dose of warfarin, liver dysfunction, alcoholism, use of another anticoagulant, use of chemotherapy, or if they do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
time to achieve the therapeutic target | 12 weeks
  time to achieve the therapeutic target during 12 weeks of treatment

SECONDARY OUTCOMES:
TTR (time in the therapeutic range) | 4 weeks and 12 weeks
  TTR mean of 4 week and 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Pereira, M.Sc, Principal Investigator — Laboratório de Genética e Cardiologia Molecular - Instituto do Coração
Locations (1):
- Heart Institute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santos PC, Marcatto LR, Duarte NE, Gadi Soares RA, Cassaro Strunz CM, Scanavacca M, Krieger JE, Pereira AC. Development of a pharmacogenetic-based warfarin dosing algorithm and its performance in Brazilian patients: highlighting the importance of population-specific calibration. Pharmacogenomics. 2015 Jul;16(8):865-76. doi: 10.2217/pgs.15.48. Epub 2015 Jun 8. PMID 26050796
- [Derived] Marcatto LR, Sacilotto L, Bueno CT, Facin M, Strunz CM, Darrieux FC, Scanavacca MI, Krieger JE, Pereira AC, Santos PC. Evaluation of a pharmacogenetic-based warfarin dosing algorithm in patients with low time in therapeutic range - study protocol for a randomized controlled trial. BMC Cardiovasc Disord. 2016 Nov 17;16(1):224. doi: 10.1186/s12872-016-0405-1. PMID 27855643